CLINICAL TRIAL: NCT06940258
Title: Efficacy of Caval Aorta Index for Fluid Optimization in Critically Ill Patients With Traumatic Brain Injury
Brief Title: Caval Aorta Index for Fluid Optimization in Traumatic Brain Injury
Acronym: CAI for fluids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Caval aorta index
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Fluid Balance
Keywords: caval aorta index; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After enrollment, patients will be randomly allocated using block into two groups of 46 patients in each group; ultrasound-guided ﬂuid management (US group) or standard care (C group)
Who Masked: Participant, Investigator
Masking Description: A vascular US expert will read the number contained in computer generated randomization software and determine group assignments. Daily; he will be responsible on prescribing of the required fluid.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other)
  Interventions: Other: control group
- ultrasound-guided caval-aorta index group (Experimental)
  Interventions: Procedure: ultrasound measurement of caval aorta index

INTERVENTIONS:
Procedure: ultrasound measurement of caval aorta index — ultrasound measurement of caval aorta index
  Arms: ultrasound-guided caval-aorta index group
Other: control group — fixed fluid prescription
  Arms: Control group

SUMMARY:
Traumatic brain injury is a leading cause of death and disability in trauma patients. As the primary injury cannot be reversed; management strategies must focus on preventing secondary injury by avoiding hypotension and hypoxia besides, maintaining appropriate cerebral perfusion pressure, which is a surrogate for cerebral blood flow.

DETAILED DESCRIPTION:
The caval aorta index is an ultrasound element, relatively new, used to assess volume status. Technically, the sonographic assessment of the inferior vena cava /aorta diameter ratio is an easy test to perform and can be performed effectively by doctors who are not experienced in the field of sonography (Kusumastuti et al .2021).

In this study; the caval aorta index will be used to guide fluid dosage in critically ill patients with traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

Traumatic brain injury diagnosed by computed tomography scan Glasgow coma score ≥ 4

Exclusion Criteria:

Inability to get consent. Pregnant and lactating women Traumatic subarachnoid hemorrhage Spinal cord injury Increased intra-abdominal pressure Abdominal aortic aneurysm Inferior vena cava (IVC) thrombus Portal hypertension Acute corpulmonale Congestive heart failure chronic hemodialysis Surgical intervention other than neurological one within the first 7 days Mechanical ventilation need during first 7 days Cardiac arrest during the first 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
fluid balance | after 96 hours from the admission
  the difference between fluid input and fluid loss

SECONDARY OUTCOMES:
Urine output | Daily for 7 weeks
  mL
Central Venous Pressure (CVP) measurements | Daily every 6 hours for 7 days
  cm H2O
Frequency and duration of hypotension | within first 7 days
  systolic blood pressure less than 90 mmhg
Glasgow Coma Scale | daily within first 7 days
  range from 3-to-15
Central capillary refill | Daily for 7 days
  seconds
incidence of pulmonary edema | Daily within first 7 days
  new B-lines in lung Ultrasound